CLINICAL TRIAL: NCT00807508
Title: The Influence of Leucine Supplementation on Body Composition and Muscle Characteristics in Healthy Elderly
Brief Title: Leucine Supplementation in Elderly Men
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Luc JC van Loon, PhD, MaastrichtUMC
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MEC 06-3-062A
Record Dates: First submitted 2008-12-11; First posted 2008-12-12 (Estimated); Last update posted 2008-12-12 (Estimated); Status verified 2008-12

CONDITIONS: Sarcopenia; Atrophy; Aging
MeSH Terms: conditions — Sarcopenia; Atrophy | interventions — Leucine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): daily leucine supplementation
  Interventions: Dietary Supplement: leucine
- 2 (Placebo Comparator): daily placebo supplementation
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: placebo — wheat meal capsules with each main meal
  Arms: 2
Dietary Supplement: leucine — daily leucine capsules with each main meal
  Arms: 1

SUMMARY:
In the present study the investigators aim to determine whether leucine supplementation can augment muscle mass and strength and improve body composition in healthy elderly men

ELIGIBILITY:
Inclusion Criteria:

* living independently

Exclusion Criteria:

* Diabetes cardiovascular disease orthopedic limitations history of resistance training in past 5 years

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-01; Primary Completion 2007-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
muscle mass and body composition | before and after 12 wk intervention

SECONDARY OUTCOMES:
muscle strength | before and after 12 wk intervention

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Centre, Maastricht, Netherlands

REFERENCES:
- [Derived] Verhoeven S, Vanschoonbeek K, Verdijk LB, Koopman R, Wodzig WK, Dendale P, van Loon LJ. Long-term leucine supplementation does not increase muscle mass or strength in healthy elderly men. Am J Clin Nutr. 2009 May;89(5):1468-75. doi: 10.3945/ajcn.2008.26668. Epub 2009 Mar 25. PMID 19321567